CLINICAL TRIAL: NCT04307901
Title: Safety Of ColoRectal Assessment and Tumor Evaluation by Colon Capsule Endoscopy
Acronym: SOCRATEC
Status: Recruiting | Type: Observational
Sponsor: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Issam al-Najami, Principal Investigator, Odense University Hospital
Other Study IDs: 20/4408
Record Dates: First submitted 2020-03-12; First posted 2020-03-13 (Actual); Last update posted 2020-05-20 (Actual); Status verified 2020-05

CONDITIONS: Colorectal Cancer; Colorectal Polyp
Keywords: colon capsule endoscopy; ct colonography; colonoscopy; endoscopy
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Endoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (3):
- Incomplete colonoscopy: Individuals referred to colon capsule endoscopy due to incomplete colonoscopy investigation.
  Interventions: Device: Colon capsule endoscopy
- Colonoscopy general anesthesia: Individuals referred to colon capsule endoscopy as alternative to colonoscopy under general anesthesia.
  Interventions: Device: Colon capsule endoscopy
- Colonoscopy declined: Individuals referred to colon capsule endoscopy after completion of bowel preparation for colonoscopy, but who have declined colonoscopy to be carried out.
  Interventions: Device: Colon capsule endoscopy

INTERVENTIONS:
Device: Colon capsule endoscopy — Endoscopy performed using PillCam2 camera capsule for oral ingestion

SUMMARY:
Following European guidelines patients undergoing colonoscopy in one of Odense University Hospitals units will now be offered a colon capsule endoscopy (CCE) in case of incomplete examinations. Patients formerly referred to colonoscopy in general anesthesia or patients who decline colonoscopy after having completed bowel preparation will also be offered a CCE. In our department we have conducted a comparison study documenting that the sensitivity of CCE is superior to CT colonography in both polyps >9 mm and polyps >5 mm, which is also supported by an Italian study. The safety and completion rate of CCE following incomplete colonoscopy is confirmed by several studies including one multicenter study and the completion rate is not significantly lower compared to other patient groups. In an incomplete colonoscopy it is always the most oral part of the colon which is not visualized, whereas in CCE, an incomplete investigation will most often have visualized the oral part. By combining incomplete colonoscopy results and incomplete CCE results we can identify patients who have had a complete colon investigation although both investigations were incomplete.

Aim: to investigate the quality of CCE and the completion rate in patients who have undergone an incomplete colonoscopy, have completed bowel preparation but declines colonoscopy or have been referred to colonoscopy in general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Incomplete colonoscopy, referral for colonoscopy under general anesthesia or declining colonoscopy after completion of bowel preparation.

Exclusion Criteria:

* Chrohn's disease with symptoms of stenosis and/or pacemaker

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adults referred to colon capsule endoscopy from the surgical department of Odense University Hospital, which signs consent form enabling us to retrieve personal data.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2020-05-01 (Actual); Primary Completion 2030-10-01 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Complete mucosal visualization combining incomplete investigations | 10 years
  By combining results from incomplete colon capsule endoscopy and incomplete colonoscopy we will identify complete combined investigations.

SECONDARY OUTCOMES:
Completion rate of colon capsule endoscopy | 2 years
  Total and subgroup completion rates of investigations
Safety of colon capsule endoscopy | 1 year
  Total and subgroup safety of investigations
Quality of colon capsule endoscopy | 1 year
  Sensitivity and specificity compared to colonoscopies
Economic evaluation | 1 year
  Economic analyses and evaluations comparing cost of investigations per patient and per case by investigation type.
Patient preference | 2 years
  Investigation of patient preferences stratified by demographic characteristics and history of endoscopic procedures

CONTACTS AND LOCATIONS:
Locations (1):
- Odense University Hospital, Svendborg, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Havshoi AV, Deding U, Jensen SS, Andersen PV, Kaalby L, Al-Najami I. Colon capsule endoscopy following incomplete colonoscopy in routine clinical settings. Surg Endosc. 2023 Apr;37(4):2749-2755. doi: 10.1007/s00464-022-09783-w. Epub 2022 Dec 5. PMID 36471059